CLINICAL TRIAL: NCT00187382
Title: Multiple Courses of Antenatal Corticosteroids for Preterm Birth Study (MACS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FRN: 38142; ISRCTN72654148
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Pregnancies at Increased Risk of Preterm Birth
Keywords: antenatal corticosteroids; preterm birth; multiple versus single doses; follow-up
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Multiple vs. single courses of antenatalcorticosteroids

SUMMARY:
In women at 26 to 30 weeks gestation and who are risk for threatened early birth, who have not had their baby by 14 or more days after being given a single course of antenatal corticosteroids (ACS), do repeated courses of ACS every 14 days until 33 weeks' gestational age lower the risk of illness or death in babies compared to repeated courses of placebo. Children are assessed at 2 years and 5 years for neurodevelopmental impairment.

DETAILED DESCRIPTION:
In women at 26 to 30 weeks gestation, who are at increased risk for preterm birth and remain undelivered 14 or more days following a single course of antenatal corticosteroids (ACS), are multiple course of ACS every 14 days until 33 weeks effective in reducing the risk of perinatal or neonatal mortality or significant neonatal morbidity, compared to placebo.

18-24 Month Follow-up: Children (18-24 months corrected gestational age) are assessed with the Bayley Scales of Infant Development (Second Edition) to determine neurodevelopmental impairment.

5 Year Follow-up (MACS-5): Children are assessed using the Child Behaviour Checklist (1 1/2 - 5) and the Behaviour Rating Inventory of Executive Function (Preschool version) to determine neurocognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Women who have previously received one completed course of ACS, at least 14 days ago and continue to be at increased risk of preterm birth
* Gestational age greater ≥ 26 weeks and gestational age < 31 weeks

Exclusion Criteria:

* Women requiring chronic doses of corticosteroids secondary to medical conditions
* Women with a contraindication to corticosteroids
* Women with clinical evidence of chorioamnionitis (temperature ≥ 38°c)
* Known lethal congenital anomaly (e.g. anencephaly)

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1858 (Actual)
Dates: Start 2001-04; Primary Completion 2007-06 (Actual); Study Completion 2011-12

PRIMARY OUTCOMES:
MACS: Perinatal or neonatal mortality or serious neonatal morbidity
MACS-5: Mortality or survival with severe neuro-morbidities at 5 years of age

SECONDARY OUTCOMES:
MACS: Death or neurologic impairment at 2 years of age
MACS-5: Measures of growth and blood pressure assessed by clinical exam
MACS-5: At Canadian sites, abnormalities in intelligence and specific cognitive skills (WPPSI-III, Beery: VMI and PPVT-III)

CONTACTS AND LOCATIONS:
Overall Officials: Kellie Murphy, M.D., Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Data Coordinating Centre, CMICR 790 Bay Street, 7th Floor, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Asztalos E, Willan A, Murphy K, Matthews S, Ohlsson A, Saigal S, Armson A, Kelly E, Delisle MF, Gafni A, Lee S, Sananes R, Rovet J, Guselle P, Amankwah K; MACS-5 Collaborative Group. Association between gestational age at birth, antenatal corticosteroids, and outcomes at 5 years: multiple courses of antenatal corticosteroids for preterm birth study at 5 years of age (MACS-5). BMC Pregnancy Childbirth. 2014 Aug 13;14:272. doi: 10.1186/1471-2393-14-272. PMID 25123162
- [Derived] Asztalos EV, Murphy KE, Willan AR, Matthews SG, Ohlsson A, Saigal S, Armson BA, Kelly EN, Delisle MF, Gafni A, Lee SK, Sananes R, Rovet J, Guselle P, Amankwah K, Saleem M, Sanchez J; MACS-5 Collaborative Group. Multiple courses of antenatal corticosteroids for preterm birth study: outcomes in children at 5 years of age (MACS-5). JAMA Pediatr. 2013 Dec;167(12):1102-10. doi: 10.1001/jamapediatrics.2013.2764. PMID 24126948
- [Derived] Murphy KE, Willan AR, Hannah ME, Ohlsson A, Kelly EN, Matthews SG, Saigal S, Asztalos E, Ross S, Delisle MF, Amankwah K, Guselle P, Gafni A, Lee SK, Armson BA; Multiple Courses of Antenatal Corticosteroids for Preterm Birth Study Collaborative Group. Effect of antenatal corticosteroids on fetal growth and gestational age at birth. Obstet Gynecol. 2012 May;119(5):917-23. doi: 10.1097/AOG.0b013e31825189dc. PMID 22525902
- [Derived] Asztalos EV, Murphy KE, Hannah ME, Willan AR, Matthews SG, Ohlsson A, Kelly EN, Saigal S, Ross S, Delisle MF, Amankwah K, Guselle P, Gafni A, Lee SK, Armson BA, Sananes R, Tomat L; Multiple Courses of Antenatal Corticosteroids for Preterm Birth Study Collaborative Group. Multiple courses of antenatal corticosteroids for preterm birth study: 2-year outcomes. Pediatrics. 2010 Nov;126(5):e1045-55. doi: 10.1542/peds.2010-0857. Epub 2010 Oct 18. PMID 20956409